CLINICAL TRIAL: NCT06605755
Title: Extended Study on the Safety and Immunogenicity of DTaP-IPV/Hib Pentavalent Vaccine in Chinese 2-month-old Infants: a Randomized, Prospective, Open Clinical Study
Brief Title: Safety and Immunogenicity of DTaP-IPV/Hib Pentavalent Vaccine in Chinese 2-month-old Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT-ZL03
Record Dates: First submitted 2024-09-04; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-08

CONDITIONS: Pertussis; Diphtheria; Tetanus; Haemophilus Influenzae Type B Infection; Polio
MeSH Terms: conditions — Whooping Cough; Diphtheria; Tetanus; Haemophilus Infections; Poliomyelitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group: 1 dose of DTaP-IPV/Hib Pentavalent Vaccine at 2, 4 and 6 months of age, and 1 dose of enhanced vaccine at 18 months of age.
  Interventions: Procedure: Different immunization regiments with DTaP-IPV/Hib Pentavalent Vaccine
- Control group (Active Comparator): Control group: 1 dose of DTaP-IPV/Hib Pentavalent Vaccine at 2, 3 and 4 months of age, and 1 dose of enhanced vaccine at 18 months of age.
  Interventions: Procedure: Different immunization regiments with DTaP-IPV/Hib Pentavalent Vaccine

INTERVENTIONS:
Procedure: Different immunization regiments with DTaP-IPV/Hib Pentavalent Vaccine — The test vaccine in this study was Pentaxim®, a pentavalent vaccine produced by Sanofi Pasteur, France.This vaccine is a combination vaccine consisting of adsorbed acellular DTP and inactivated polio vaccine (DTaP-IPV) and Haemophilus influenzae type b conjugate vaccine (Hib).
  1. Intervention group: 1 dose of experimental vaccine at 2, 4 and 6 months of age, and 1 dose of enhanced vaccine at 18 months of age.
  2. Control group: 1 dose of experimental vaccine at 2, 3 and 4 months of age, and 1 dose of enhanced vaccine at 18 months of age.

SUMMARY:
The main purpose of this study is to evaluate immune persistence at 30 and 36 Months of Age and Pertussis Breakthrough Infections between 19 and 36 Months of Age following two regiments of DTaP-IPV/Hib Pentavalent Vaccine in Healthy 2-Month-Old Infants and Children in China.

DETAILED DESCRIPTION:
This study was based on the DTaP-IPV/Hib Pentavalent Vaccine Basic Immunization Strategy Optimization Study Cohort ("Pentavalent Vaccine Cohort") and the Epidemiological Investigation of Carrying Status of Pathogens Causing Acute Respiratory Infections (ARIs) in Infants and Young Children Cohort ("Pathogen Surveillance Cohort").

DTaP-IPV/Hib vaccine basic immunization strategy optimization study is a single-center, randomized, prospective and open clinical trial. The study was designed for two groups: 2, 3, 4, 18 months of age (control group) and 2, 4, 6, 18 months of age (intervention group). Subjects were randomly assigned to two groups according to the principle of informed consent. Collect basic demographic information of children and their families. The control group received 3 doses of acellular DPT vaccine at 2, 3 and 4 months of age respectively, and 1 dose at 18 months of age; The intervention group received 3 doses of acellular DPT vaccine at 2, 4 and 6 months of age respectively, and 1 dose at 18 months of age. The immunogenicity and safety were observed before and after 28 days of 3 doses of basal immunization, and after 28 days of enhanced immunization at 18 months of age.

The pathogen surveillance team included 2-month-old infants and caregivers with whom they shared a life history. After informed consent, the researchers followed up the subjects from 2 months of age to 19 months of age. The main contents of the visit are sample collection and unified questionnaire survey.

On the basis of the surveillance of ARI aged 2 to 19 months, follow-up was conducted for 17 months. During the follow-up period, ARI telephone visit was conducted twice a week. After ARI was found, pathogen sampling and testing were conducted for them (participants and their caregivers) to monitor the emergence of pertussis infection. Blood samples and throat swabs were collected at 30 and 36 months of age (caregivers were also required to take simultaneous samples), and penta vaccine immunity persistence was observed and multiple respiratory pathogens were monitored.

ELIGIBILITY:
Inclusion Criteria:

- (1)Received 4 doses of DTaP-IPV/Hib pentavalent vaccines (2) Obtained consent from the participant's caregiver and sign an informed consent form

Exclusion Criteria:

-(1) Diagnosed by a physician with a coagulation abnormality (e.g., coagulation factor deficiency, coagulopathy, platelet abnormality) (2) Any other factor considered to make participation in the trial unsuitable.

Ages: 19 Months to 22 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 785 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Anti-pertussis toxin, anti-pertussis filamentous hemagglutinin, anti-pertussis adhesin, anti-pertussis FIM2, anti-pertussis FIM3 .Anti-diphtheria, anti-tetanus, anti-HIB PRP and anti-type 1, 2 and 3 poliomyelitis antibody levels . | 30 months of age
  Measure antibody levels
Anti-pertussis toxin, anti-pertussis filamentous hemagglutinin, anti-pertussis adhesin, anti-pertussis FIM2, anti-pertussis FIM3 .Anti-diphtheria, anti-tetanus, anti-HIB PRP and anti-type 1, 2 and 3 poliomyelitis antibody levels . | 36 months of age
  Measure antibody levels

SECONDARY OUTCOMES:
The positive rate of anti-pertussis toxin, anti-pertussis filamentous hemagglutinin , anti-pertussis adherin, anti-pertussis FIM2, anti-pertussis FIM3 ,anti-diphtheria , anti-tetanus , anti-HIB PRP and anti-type 1, 2, 3 poliomyelitis antibody | 30 months of age
  Measure positive rate of antibody and the growth multiple of GMC
The positive rate of anti-pertussis toxin, anti-pertussis filamentous hemagglutinin , anti-pertussis adherin, anti-pertussis FIM2, anti-pertussis FIM3 ,anti-diphtheria , anti-tetanus , anti-HIB PRP and anti-type 1, 2, 3 poliomyelitis antibody | 36 months of age
  Measure positive rate of antibody and the growth multiple of GMC
To evaluate the pathogen detection rates of ARI in 2-month-old healthy infants in China after different DTaP-IPV/Hib vaccination programs during 19-36 months of age. | 19-36 months of age
  The pathogen detection rate was calculated.
To evaluate the pertussis breakthrough infection rate in healthy infants and young children aged 19 to 36 months after receiving DTaP-IPV/Hib vaccine. | 19-36 months of age
  To evaluate the pertussis breakthrough infection rate.

CONTACTS AND LOCATIONS:
Overall Officials: jingxin42102209@126.com Li, Study Director — Jingsu Provincial Centre of Disease Control and Prevention
Locations (1):
- Jingsu Provincial Centre of Disease Control and Prevention, Nanjing, Jiangsu, China